CLINICAL TRIAL: NCT04999098
Title: Randomized, Controlled, 3-arm, Open, Prospective Clinical Trial to Assess Antiviral Properties of Echinacea Reducing Oropharyngeal Concentration and Infectivity of SARS-CoV-2: The Shedding Study
Brief Title: Echinaforce COVID-19 Shedding Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: A. Vogel AG (Industry)
Collaborators: Clinical Research Centre CONVEX (Unknown); Biodome Clinical (Unknown); MediStat Ltd. (Unknown); Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5'000'820
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Respiratory Infection; SARS-CoV2 Infection
Keywords: SARS-CoV2 infectivity; Viral load reduction; antiviral treatment; Oropharynx; Throat
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, 3-armed, parallel, active-treatment controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- treatment group 1: Echinaforce Forte (EFF) Tablets (chewed) (Active Comparator): 1st arm (EFF group): Slowly sucking 1 Echinaforce Forte tablet (1 tablet: 1'200mg EF) until dissolution "Dose 1". Another 2 X 1 EF Forte tablets (total of 2 tablets: 2'400 mg EF) is taken one-by-one "Dose 2" after swab sampling, which is repeated after complete dissolution of the second dose of EF Forte tablets.
  Interventions: Drug: Echinaforce Forte tablets
- treatment gorup 2: Echinaforce Chewable (EFC) Tablets (chewed) (Active Comparator): 2nd arm (EFC group): Slowly sucking 1 x 3 Echinaforce Chewable tablets (total 3 tablets: 1'200mg EF) until dissolution "Dose 1". Another dose of 2 x 2 & 1 x 3 EF Chewable tablets (total 7 tablets: 2'800mg EF) are slowly sucked "Dose 2" after swab sampling, which is repeated after complete dissolution of the second dose of EF Chewable tablets.
  Interventions: Drug: Echinaforce Chewable tablets
- treatment group 3: Echinaforce Tincture (EFT, gargling) (Active Comparator): 3rd arm (EFT group): Gargling of 2 x 19 drops of Echinaforce tincture (1'200 mg EF) is diluted in 2 x35 mL water "Dose 1". Another dose of 3 x 30 drops of Echinaforce tincture (2'800 mg EF) diluted in 3 x35 mL water for 15 sec each "Dose 2", gargled for 15 sec and swallowed after swab sampling, which is repeated after gargling of the second dose of EF Tincture.
  Interventions: Drug: Echinaforce tincture

INTERVENTIONS:
Drug: Echinaforce Forte tablets — Tincture of fresh Echinacea purpurea (L) MOENCH: Herba rec. T. aerial part DER = 1:12-13 (Drug to extraction solvent ratio) extraction solvent = ethanol 65.1 % (V/V) = 57.3 % (m/m)* with an approx. dry plant equivalent of 32 mg per tablet Dry weight content in 1 tablet: 5.9 mg
  Echinacea purpurea: (L) MOENCH: Radix rec. root part DER = 1:11-12 (Drug to extraction solvent ratio) extraction solvent = ethanol 65.1 % (V/V) = 57.3 % (m/m)* with an approx. dry plant equivalent of 1.8 mg per tablet Dry weight content in1 tablet: 0.3 mg
  the tablet contain additional excipients
  Arms: treatment group 1: Echinaforce Forte (EFF) Tablets (chewed)
Drug: Echinaforce Chewable tablets — Tincture of fresh Echinacea purpurea (L) MOENCH: Herba rec. T. aerial part DER = 1:12-13 (Drug to extraction solvent ratio) extraction solvent = ethanol 65.1 % (V/V) = 57.3 % (m/m)* with an approx. dry plant equivalent of 32 mg per tablet Dry weight content in 1 tablet: 5.9 mg
  Echinacea purpurea: (L) MOENCH: Radix rec. root part DER = 1:11-12 (Drug to extraction solvent ratio) extraction solvent = ethanol 65.1 % (V/V) = 57.3 % (m/m)* with an approx. dry plant equivalent of 1.8 mg per tablet Dry weight content in1 tablet: 0.3 mg
  The tablets contain additional excipients
  Arms: treatment gorup 2: Echinaforce Chewable (EFC) Tablets (chewed)
Drug: Echinaforce tincture — Tincture of fresh Echinacea purpurea (L) MOENCH: Herba rec. T. aerial part DER = 1:12-13 (Drug to extraction solvent ratio) extraction solvent = ethanol 65.1 % (V/V) = 57.3 % (m/m)
  Echinacea purpurea: (L) MOENCH: Radix rec. root part DER = 1:11-12 (Drug to extraction solvent ratio) extraction solvent = ethanol 65.1 % (V/V) = 57.3 % (m/m)
  Other Names: Echinaforce drops
  Arms: treatment group 3: Echinaforce Tincture (EFT, gargling)

SUMMARY:
Respiratory viruses pose a permanent threat to humans and society as demonstrated by the current Covid-19 pandemic. Novel drugs and vaccines provide a means for controlling illness. Infections and symptomatic presentation of illness may be reduced, but it remains to be determined to which extent viral shedding and transmission (e.g. by silent transmitters) can be controlled. Lack of such activity may result in continuing viral spread by assumed healthy but asymptomatic spreaders. Echinacea is an established and readily-accessible product with demonstrated in vitro antiviral activity (including coronaviruses). This study aims to estimate the potential of different Echinacea formulations (head-to-head) to reduce concentration infectivity and shedding of SARS-CoV-2 under in vivo conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 75 years.
* Written informed consent.
* Ability and willingness to give oropharyngeal swab samples.
* Positive pre-screening SARS-CoV-2 RT-PCR virus test with an above threshold viral load as per qPCR (Cq ≤ 27).

Exclusion Criteria:

* ≥76 years
* <12 years.
* Participation in another clinical study in the past 30 days or planned during study conduct.
* Severe COVID19
* Intake of antimicrobial, antiviral, immune suppressive substances.
* Surgical intervention in the 3 months prior enrolment
* Known diabetes mellitus.
* Known and medicated atopy or asthma.
* Cystic Fibrosis, bronchopulmonary dysfunction, COPD.
* Known immune system disorders and degenerative disorders (autoimmune disorders, AIDS, leukemia, lymphoma, myeloma).
* Known metabolic or resorption disorders.
* Known liver or kidney illnesses (chronic hepatitis, liver cirrhosis, chronic kidney insufficiency).
* Serious health conditions (limited general condition, auto-immune diseases, tumorous diseases, neurological disorders or serious Covid-19)
* Known allergies to plants of the compositae family (e.g. chamomile or dandelion) or to one of the compounds in the investigational product
* Known pregnancy.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Absolute and relative differences in Cq values (qPCR) comparing pre- and post EF treatment including all formulations combined. | 2 hours
  The average Cq values as per qPCR analysis by means of qPCR values prior any treatment (samples A1 & B1) in comparison to post EF treatment. Oropharyngeal (OP) Swab samples are taken by using validated swab sticks (Eswab 480CE LQ Amies with Reg. Nylon Flocked applicator, COPAN Int.) and presence of viral RNA/DNA determined by using the qPCR SARS-CoV2 panel. The analysis is done by a two-sided t-test

SECONDARY OUTCOMES:
Absolute and relative viral loads comparing pre- and post EF treatment and in cross comparison of the respective EF-formulations | 2 hours
  The viral load reduction as per averages of Cq values and/or genomic read depths (optional) prior any treatment (samples A1 & B1) in comparison to post EF treatment and/or in cross-comparison with the respective time point and/or formulation. Oropharyngeal (OP) Swab samples are taken by using validated swab sticks (Eswab 480CE LQ Amies with Reg. Nylon Flocked applicator, COPAN Int.) and presence and quantity of viral RNA/DNA determined by using the qPCR SARS-CoV2 panel. The viral genomic material is optionally quantified by genomic read depth as per next generation sequencing (NGS). The analysis is done by a two-sided t-test for comparing pre- and post-treatment and ANOVA for cross-comparisons between groups
Absolute and relative tissue infective dose (TCID) of recovered life viruses comparing pre- and post EF treatment results and/or in cross-comparison of the respective EF formulations. | 2 hours
  Residual tissue culture infectious dose per time point: prior any treatment (pre-treatment samples A1 & B1), to post EF treatment and/or in cross-comparison with the respective time point and/or formulation. The analysis is done by a two-sided t-test for comparing pre- and post-treatment and ANOVA for cross-comparisons between groups
Incidence of Treatment responders falling below limit of detection/ threshold value under treatment | 2 hours
  The number of subjects per time point that become qPCR negative as per RT-PCR test results and/or reached below threshold genomic read depth value (optional) as per NGS-read out and reach a below threshold residual infectivity as per TCID test result are determined prior and post EF treatment and in cross-comparison of the respective EF formulations. The analysis is done by non-parametric chi-square endpoint analysis].
Incidence of SARS-CoV-2 VOC (variant of concerns) | 2 hours
  Absolute and relative frequencies of SARS-CoV2 VOCs is as per identification by optional whole-genome next generation sequencing and automated database annotation to known and unknown SARS-CoV2 strains on pre-treatment samples A1 & A2. The analysis is done by non-parametric chi-square endpoint analysis
Frequency of concomitant medication/therapies | 3 days
  The use of any concomitant medication and/or application of therapies in patients is assessed during home visit as per eCRF entries. The analysis is done by non-parametric chi-square endpoint analysis
Frequency of intake of pre-treatment, Beverage and food-intake prior therapy start. | 3 days
  The use of any relevant pre-treatment, beverage and food consumption in patients is assessed during home visit as per eCRF entries. Any such intake in any case shall be recorded in the eCRF
Frequency of vaccination | 2 hours
  The vaccine or prevention status of patients is assessed during home visit as per eCRF entries. Patients are asked if they have obtained SARS-CoV2 vaccination in the past. If yes, which one incl. full product name, number of vaccination shots, time point of vaccination?
Tolerability in view of subjects after treatment. | 2 hours
  The treatment tolerability per corresponding study product is assessed by subjects after completion of all study procedures during home visit as per eCRF entries by asking the question how they rate the tolerability of their corresponding study product on a scale: bad = 0, average = 1, good = 2, very good = 3). The analysis is done by Mantel-Haenszel test].
Tolerability in view of Investigators after treatment. | 2 hours
  The treatment tolerability per corresponding study product is assessed by the study investigators after completion of all study procedures during home visit as per eCRF entries by asking the question how they rate the tolerability in the subject of the corresponding study product on a scale: bad = 0, average = 1, good = 2, very good = 3). The analysis is done by Mantel-Haenszel test].
Incidence and severity of other symptoms (S/AEs). | 2 hours
  S)AE, occurring during home visits are being detected as per e-CRF entries during home visit after study inclusion. Such events are additionally assessed after termination of the study in the form of a compiled safety report. Absolute and relative frequencies are analysed descriptively by non-parametric Fishers-exact/Chi2 test]

CONTACTS AND LOCATIONS:
Locations (1):
- Diagnostics and Consultation Center Convex EOOD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan yet